CLINICAL TRIAL: NCT01099618
Title: Ketosis-Prone Diabetes in African Americans: Predictive Markers, Underlying Mechanisms, and Treatment Outcomes: The Effects of Metformin vs. Sitagliptin on Beta-Cell Preservation in Obese Subjects With Ketosis-Prone Type 2 Diabetes Mellitus
Brief Title: Ketosis-Prone Diabetes Mellitus (KPDM): Metformin Versus Sitagliptin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dawn Smiley MD (Other)
Responsible Party: Sponsor-Investigator, Dawn Smiley MD, Principal Investigator, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00026272
Record Dates: First submitted 2010-03-15; First posted 2010-04-07 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Ketosis Prone Diabetes; Diabetes Ketoacidosis; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin (Active Comparator): All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA (N=24) and obese subjects with hyperglycemia without ketoacidosis (n=24) will be equally randomized to receive metformin (MET) 1000 mg (n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  Interventions: Drug: metformin
- Sitagliptin (Active Comparator): All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000 mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA (N=24) and obese subjects with hyperglycemia without ketoacidosis (n=24) will be equally randomized to receive metformin (MET) 1000 mg (n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000 mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA (N=24) and obese subjects with hyperglycemia without ketoacidosis (n=24) will be equally randomized to receive metformin (MET) 1000 mg(n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metformin — The study subject will receive metformin (MET) 1000 mg tablet once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
  Other Names: Glucophage
  Arms: Metformin
Drug: placebo — The study subject will receive a placebo tablet once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
  Arms: Placebo
Drug: Sitagliptin — The study subject will receive a sitagliptin 100mg once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
  Other Names: Januvia
  Arms: Sitagliptin

SUMMARY:
The study intends on enrolling 48 subjects with diabetes. Diabetic subjects that no longer need insulin will be randomly placed (like the flip of a coin) on a diabetes pill called metformin, a diabetes pill called sitagliptin or a placebo pill (a pill without active medication). Subjects on pills will be followed for 3½ years and undergo blood tests at specified intervals to assess their ability to make insulin. These studies will allow a better understanding of the factors that lead to high blood sugar in patients with ketosis-prone diabetes mellitus (KPDM) and direct the best diabetes treatment for this patient population.

Hypothesis: Metformin therapy or sitagliptin therapy compared to placebo, will improve β-cell function, insulin sensitivity, and allow for a longer period of time prior to encountering an insulin-deficient relapse after discontinuation of insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. All newly diagnosed overweight/obese (BMI >/=28 kg/m2) African-American patients with new-onset DKA and/or severe hyperglycemia and without apparent precipitating cause will be considered for inclusion into the study. The diagnosis of DKA will be established by standard criteria (blood glucose > 250 mg/dL, pH < 7.3, HCO3 < 18 mmol/L, increased anion gap).
2. The hyperglycemic group will include patients with an admission plasma glucose > 400 mg/dL but without the presence of metabolic acidosis or ketosis.

Exclusion Criteria:

1. significant medical or surgical illness, including but not limited to myocardial ischemia, congestive heart failure, chronic renal insufficiency, liver failure, and infectious processes;
2. recognized or suspected endocrine disorders associated with increased insulin resistance, such as hypercortisolism, acromegaly, or hyperthyroidism;
3. bleeding disorders, thrombocytopenia, or abnormalities in coagulation studies;
4. pregnancy,
5. have an allergy to any component of metformin or sitagliptin.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn D. Smiley, MD, Principal Investigator — Emory School of Medicine
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Vellanki P, Stefanovski D, Anzola II, Smiley DD, Peng L, Umpierrez GE. Long-term changes in carbohydrate tolerance, insulin secretion and action in African-American patients with obesity and history of hyperglycemic crises. BMJ Open Diabetes Res Care. 2020 May;8(1):e001062. doi: 10.1136/bmjdrc-2019-001062. PMID 32475838
- [Derived] Vellanki P, Smiley DD, Stefanovski D, Anzola I, Duan W, Hudson M, Peng L, Pasquel FJ, Umpierrez GE. Randomized Controlled Study of Metformin and Sitagliptin on Long-term Normoglycemia Remission in African American Patients With Hyperglycemic Crises. Diabetes Care. 2016 Nov;39(11):1948-1955. doi: 10.2337/dc16-0406. Epub 2016 Aug 29. PMID 27573938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: new onset type 2 diabetes with BG > 400 or with DKA
Period: Overall Study
Arm/Group | Metformin | Sitagliptin | Placebo
Started | 17 | 16 | 15
Completed | 17 | 16 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: AA patient with new-onset DM presenting with BG > 400 or DKA
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 15 | 48
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9) | 50 (11) | 48 (7) | 48 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 7 | 18
  Male | 11 | 11 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 16 | 15 | 48
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Length of Remission
Description: For those patients that are able to discontinue insulin therapy at or <12 weeks, how long were they able to well controlled with an A1c <7% on the agent that they were randomized to.
Time Frame: 3 years
Measure: Median (Full Range); unit: days
Arm/Group | Metformin | Sitagliptin | Placebo
Number analyzed (Participants) | 17 | 16 | 15
days | 472 [95 to 1189] | 589 [89 to 977] | 111 [43 to 1015]

ADVERSE EVENTS:
Time Frame: 3 years, during the time of the study
Groups:
- Metformin: All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA and without ketoacidosis will be randomized to receive metformin (MET) 1000 mg (n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  metformin: The study subject will receive metformin (MET) 1000 mg tablet once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
- Sitagliptin: All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000 mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA and without ketoacidosis will be randomized to receive metformin (MET) 1000 mg (n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  Sitagliptin: The study subject will receive a sitagliptin 100mg once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
- Placebo: All newly diagnosed subjects with KPDM that are able to discontinue insulin after 12 weeks or less will be randomized in double-blind fashion to receive either metformin 1000 mg, sitagliptin 100mg or placebo once daily. Subjects that do not achieve remission will continue to receive insulin therapy and will discontinue the protocol. A total of 48 obese subjects with DKA and without ketoacidosis will be randomized to receive metformin (MET) 1000 mg(n=16), sitagliptin (SIT) 100mg (n=16) or placebo (n=16).
  placebo: The study subject will receive a placebo tablet once a day as long as the patient maintains near-normoglycemic remission (BG < 130mg/dL and A1c <7%) during the 3-year follow-up period.
Arm/Group | Metformin | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/17 | 1/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=17) | Sitagliptin (N=16) | Placebo (N=15)
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) — loose stool after starting the medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes